CLINICAL TRIAL: NCT01614145
Title: Diagnostic Study Evaluating the Performance of an Aspergillus-specific Nested PCR Assay in Cerebrospinal Fluid Samples of Immunocompromised Patients for Detection of Central Nervous System Aspergillosis
Brief Title: Diagnostic Performance of an Aspergillus-specific Nested PCR Assay in Cerebrospinal Fluid Samples
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dieter Buchheidt, Prof. Dr., Heidelberg University
Other Study IDs: CSF Aspergillus PCR
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Focus: Immunocompromised Individuals at High Risk of Aqcuiring Invasive Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Aspergillus DNA samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Proven/probable CNS IA: Immunocompromised patients with proven/probable invasive CNS Aspergillosis based on modified criteria by the EORTC/MSG
- Possible/No CNS IA: Immunocompromised patients with possible/NoIA invasive CNS Aspergillosis based on modified criteria by the EORTC/MSG

SUMMARY:
Multicentre, diagnostic study evaluating the performance of an aspergillus-specific PCR in cerebrospinal fluid samples of immunocompromised patients for identification of central nervous system aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

* Host factors
* Informed consent

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Immunocompromised patients at risk for invasive aspergillosis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-09; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Test sensitivity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Buchheidt, MD, Principal Investigator — Germany: Mannheim University Hospital, University of Heidelberg
Locations (3):
- Germany (3):
  - Freiburg University Hospital, Freiburg im Breisgau, Baden-Würrtemberg
  - Mannheim University Hospital, Mannheim, Baden-Würrtemberg
  - Frankfurt (Oder) General Hospital, Frankfurt (Oder), Brandenburg